CLINICAL TRIAL: NCT06083506
Title: Immediate Loading of 4 Guided Implants Supporting a Maxillary Overdenture Using a Novaloc TiN Retention System: Open Ended Prospective Study
Brief Title: Immediate Loading of 4 Guided Implants Supporting a Maxillary Overdenture Using a Novaloc TiN Retention System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: West Virginia University (Other)
Collaborators: Institut Straumann AG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1801929813
Record Dates: First submitted 2023-10-03; First posted 2023-10-16 (Actual); Results first posted 2025-07-20 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Immediate Dental Implant Loading; Denture, Complete

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- NOVALOC TiN (Other): Each subject will receive 4 implants. Implants will be placed flapless using a guided surgical protocol and will be immediately loaded by means of a NOVALOC TiN retained maxillary overdenture.
  Interventions: Device: NOVALOC TiN retained maxillary overdenture

INTERVENTIONS:
Device: NOVALOC TiN retained maxillary overdenture — 4 implants immediately loaded by means of a NOVALOC TiN retained maxillary overdenture

SUMMARY:
Complete dentures represent the traditional dental treatment for patients without teeth. However, retention and stability of this type of denture are often lacking, so dental implants are indicated in order to improve the stability of the denture, along with the satisfaction of the patient. Usually, the dental implants are inserted and then a period of 3-6 months is waited before any denture is connected to them. Recent studies have demonstrated that connecting the lower denture to the implants immediately after the implant placement, leads to an improvement in the result, with a social and psychological benefit for the patient. Therefore, the aim of this research project is to evaluate the application of the immediate connections of the implants for the upper dentures. 15-40 patients wearing an upper denture will receive 4 dental implants and the denture will be immediately connected. To simplify the surgical procedure, the implants will be placed without exposing the bone. This surgical technique is called guided surgery. Secondary objective of this research project will be the evaluation of the precision of the implant positioning, using this specific technique. The patients will be followed up for 12 months, for the implant and denture evaluation, as well as the evaluation of patient satisfaction and impact on quality of life through questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous maxilla
* The implant site has to be healed for at least 4 months after extraction
* Wearing complete dentures deemed adequate
* Orthopantomogram available (OPT)
* Adequate amount of bone at least at the 2nd premolar position to house a 3.75 x 10 mm implant
* No bone grafting required
* Implant IT ≥ 20 N/cm

Exclusion Criteria:

* Conditions requiring chronic routine prophylactic use of antibiotics
* Conditions requiring prolonged use of steroids
* History of leukocyte dysfunction and deficiencies
* Bleeding disorders
* History of neoplastic disease requiring use of radiation or chemotherapy
* Metabolic bone disorders
* Uncontrolled endocrine disorder
* Use of any investigational drug or device within the 30-day period prior to implant surgery
* Smoking more than 10 cigarettes a day
* Alcoholism or drug abuse
* Patient infected with HIV
* Condition or circumstances, in the opinion of the investigator, which would prevent completion of study participation or interfere with analysis of study results, such as history of non-compliance, unreliability.

Local exclusion criteria:

* Local inflammation including untreated periodontitis
* Mucosal disease such as erosive lichen planus
* History of local irradiation therapy
* Osseous lesion
* Severe bruxism and clenching habits
* Active infection with suppuration or fistula track
* Persistent intraoral infection
* Lack of primary stability <20Ncm. In this instance, the patient must be withdrawn and treated according to the standard protocol.
* Inadequate oral hygiene or unmotivated home care.
* Bone grafting
* Inadequate bone volume for implants insertion as measured on the per-treatment CBCT.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2023-05-15 (Actual); Study Completion 2023-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Arif Salman, BDS, MDSc, Principal Investigator — West Virginia University
Locations (1):
- West Virginia University, Morgantown, West Virginia, United States

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Implants
Groups:
- NOVALOC TiN: Implants will be placed flapless using a guided surgical protocol and will be immediately loaded by means of a NOVALOC TiN retained maxillary overdenture.
Period: Overall Study
Arm/Group | NOVALOC TiN
Started | 17; 68 Implants
Completed | 14; 56 Implants
Not Completed | 3; 12 Implants
Not completed — Physician Decision | 2
Not completed — Lack of Efficacy | 1

BASELINE CHARACTERISTICS:
Arm/Group | NOVALOC TiN
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.2 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 12
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetics [Count of Participants; unit: Participants] | 4
Tobacco Use Status [Count of Participants; unit: Participants] | 1

OUTCOME MEASURES:

1. Primary Outcome: Radiographic Bone Level (RBL) Change
Description: RBL change will be measured in mm on standardized periapical radiographs. The distance between the implant platform and the most coronal level of the bone deemed to be in contact with the implant surface will be evaluated. Mesial and distal bone height measurements will be averaged for each implant. The measurements of the bone level at implant placement will be considered as baseline. The RBL change will be calculated in comparison with the baseline value.
Time Frame: Baseline to 6 months post implant
Measure: Mean (Standard Deviation); unit: millimeters (mm)
Units Other Than Participants: Implants
Arm/Group | NOVALOC TiN
Number analyzed (Participants) | 14
Number analyzed (Implants) | 56
millimeters (mm) | 0.14 (0.36)

2. Primary Outcome: Radiographic Bone Level (RBL) Change
Description: as for outcome 1
Time Frame: Baseline to 12 months post implant
Measure: Mean (Standard Error); unit: millimeters (mm)
Units Other Than Participants: Implants
Arm/Group | NOVALOC TiN
Number analyzed (Participants) | 14
Number analyzed (Implants) | 56
millimeters (mm) | 0.31 (0.73)

ADVERSE EVENTS:
Time Frame: 12 Months
Arm/Group | NOVALOC TiN
All-Cause Mortality (participants affected / at risk) | 0/14
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 0/14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT06083506/Prot_SAP_000.pdf
  • Informed Consent Form (2021-12-15): https://cdn.clinicaltrials.gov/large-docs/06/NCT06083506/ICF_002.pdf